CLINICAL TRIAL: NCT02039128
Title: A Double-blind, Randomized, Placebo-controlled Study to Assess Changes in the Omega-3 Index in Erythrocytes After Twelve Weeks of Daily Intake of SuperbaTM Krill Oil or Fish Oil
Brief Title: KOmparison Study KOmparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aker BioMarine Human Ingredients AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: BTS743/13 // AKBM109H
Record Dates: First submitted 2014-01-07; First posted 2014-01-17 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Krill oil (Experimental): 1 gram per day in 12 weeks
  Interventions: Dietary Supplement: Krill oil or Fish oil
- Fish oil (Active Comparator): 1 gram per day in 12 weeks
  Interventions: Dietary Supplement: Krill oil or Fish oil
- Placebo (Placebo Comparator): 1 gram per day in 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Krill oil or Fish oil
  Arms: Fish oil; Krill oil
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
In this double blind, placebo controlled, parallel group study, the relative uptake of 1g/d krill oil in comparison to 1g/d fish oil in healthy female and male adults will be assessed.

Primary objective is to determine if a 12 week supplementation with krill oil increases tissue levels in erythrocytes (omega-3 index) significantly more than fish oil after dose adjustments to EPA and DHA levels.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Be able to communicate well with the Investigator, to understand and comply with the requirements of the study, and be judged suitable for the study in the opinion of the Investigator
* Be in general good health with no existing co-morbidities
* Be aged between 20 and 50 years
* Both genders allowed (at least 40% of each gender to be recruited into the study)
* Have a body mass index (BMI) between 19 and 30 kg/m² (extremes included)
* Have a omega-3 index in erythrocytes of <6.2% at screening
* Have clinically normal findings for haematology and clinical chemistry (or clinically insignificant, if value is outside of the normal range)
* Be willing to maintain dietary habits and physical activity levels throughout the trial period (next 12 weeks)
* Have a low habitual consumption of fatty fish and seafood, defined as a frequency of twice per month or less (a list of fish and seafood considered to be fatty is provided to volunteers)
* Be willing to avoid all fish and seafood meals in the 3 days before each scheduled clinic visit
* Be willing to avoid alcohol in the 24 hours before each scheduled clinic visit
* Be willing to avoid sportive activity in the 24 hours before each scheduled clinic visit
* Be willing to complete questionnaires, records and diaries associated with the study

Exclusion Criteria:

* Smoking
* Diseases or disorders that include: Rheumatoid arthritis, chronic serious illness, cardiovascular problems, liver and kidney disease, diabetes, endocrine or metabolic disease, inflammatory bowel disease, pancreatitis, gallbladder or biliary disease, neurological or psychological disease, bleeding disorders, experiences platelet abnormalities, gastrointestinal disorders that could interfere with fat absorption, acute and history of cancer, HIV, hepatitis B or C, an intention to lose weight
* Pregnant or nursing women or women of child-bearing potential whose urinary pregnancy test at screening is positive
* Postmenopausal women
* Known allergy to crustaceans (shellfish) or fish
* Known alcohol or drug abuse within the previous year of screening
* More than 20 alcohol Units per week
* Clinically significant illness within 3 days prior to dosing (fever; inability to work etc.)
* Donation of blood or similar blood loss within the previous 30 days before screening
* Participation in a clinical trial with an investigational product within 90 days before screening
* Present or recent use (within 3 months of screening) of any medication which is a known lipid modifying agent
* Present or recent use (within 3 months of screening) of dietary supplements that affect the level of blood cholesterol and triglycerides, such as fish oil supplements, niacin, etc
* Patients with known coagulopathy or receiving anticoagulant therapy or co-morbidity that would interfere with the study results
* Frequency of fatty fish and/or seafood consumption is greater than twice per month
* Present or recent use (within 3 months of screening) of any long-chain omega-3 or omega-6 fatty acid supplement

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in relative amount of EPA and DHA in erythrocytes | Baseline to Week 12

SECONDARY OUTCOMES:
Number of participants with Adverse Events as a Measure of Safety and Tolerability | Baseline to Week 12
Change in relative amount of EPA and DHA in erythrocytes | Baseline to Week 6
Blood lipid status | Baseline to Week 12
Quality of Life | Baseline to week 12
Mood Scores by a Likert Scale | Baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Trygve Bergeland, PhD, Study Director — Aker BioMarine Human Ingredients AS
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany